CLINICAL TRIAL: NCT06527807
Title: Clinical Characteristics and Prognosis of Acute Stroke in Pregnancy and Puerperium: A Retrospective, Observational, Nationwide, Multicenter Study
Brief Title: Clinical Characteristics and Prognosis of Acute Stroke in Pregnancy and Puerperium
Acronym: ASPP
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Affiliated Hospital of Jiangnan University (Other); Affiliated Hospital of Nantong University (Other); Baotou Central Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Jiangyin People's Hospital (Other); Qianfoshan Hospital (Other); RenJi Hospital (Other); Second Affiliated Hospital of Soochow University (Other); Second Hospital of Shanxi Medical University (Other); Shanxi Bethune Hospital (Other); Shenzhen Second People's Hospital (Other); The Affiliated Hospital of Qingdao University (Other); The First Affiliated Hospital of Nanchang University (Other); The First Affiliated Hospital of University of Science and Technology of China (Other); The First Affiliated Hospital of Zhengzhou University (Other); The Second Affiliated Hospital of Hainan Medical University (Other); Lanzhou University Second Hospital (Other); Tianjin Huanhu Hospital (Other); Tianjin Medical University General Hospital (Other); West China Hospital (Other); Xiangya Hospital of Central South University (Other); Xinxiang Central Hospital (Other); Zhejiang Provincial People's Hospital (Other); Binzhou Medical University (Other); Chongqing Medical University (Other); Tibetan Second People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: KY2024-180-01
Record Dates: First submitted 2024-07-21; First posted 2024-07-30 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Pregnancy-associated or Puerperium-associated Acute Stroke
Keywords: Acute stroke; Pregnancy; Puerperium; Clinical characteristics; Prognosis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ASPP: Patients with acute stroke in pregnancy or puerperium
- Pregnant/Puerperal Non-Stroke: Pregnant or puerperal participants without any history of stroke
- Non-Pregnant Stroke: Non-pregnant or non-puerperal participants with a recent acute stroke event

SUMMARY:
The objectives of this study are: (1) to describe the detailed clinical characteristics and prognosis of ASPP patients in order to explore the risk factors of ASPP, and to compare the short-term and long-term functional recovery outcomes between them and their controls; (2) to evaluate the risk of recurrent stroke, particularly during subsequent pregnancies, in ASPP patients; (3) to assess the short-term and long-term outcomes of their offsprings and their future development status.

This study is divided into three parts. The first part is a case-control study to explore the risk factors of ASPP and the predictors of the prognosis of ASPP patients. The second part is a cohort study to evaluate the impact of ASPP on the risk of recurrent stroke. The third part is a cohort study to assess the impact of ASPP on the short-term and long-term outcomes of their offsprings by comparing the offsprings of ASPP patients with the offsprings of non-ASPP participants.

ELIGIBILITY:
1. Case-control Study and Cohort Study on Recurrent Stroke Risk:

Inclusion Criteria:

1. Female patients ≥18 years of age;
2. Patients or their legally acceptable representatives or relatives agree to collect personal information for this study and sign an oral or online written informed consent.

Exclusion Criteria:

1. Patients or their legally acceptable representatives or relatives refuse follow-up;
2. Patients missing critical baseline demographic, clinical or neuroimaging data.

2. Cohort Study on Offspring Outcomes:

Inclusion Criteria:

1. Female patients ≥18 years of age;
2. Patients in pregnancy or within 6 weeks postpartum;
3. Patients or their legally acceptable representatives or relatives agree to collect personal information for this study and sign an oral or online written informed consent.

Exclusion Criteria:

1. Patients or their legally acceptable representatives or relatives refuse follow-up;
2. Patients missing critical baseline demographic, clinical or neuroimaging data;
3. Patients whose offsprings have congenital malformation or inborn error of metabolism;
4. Patients with complications which may affect cerebral blood flow supply, such as amniotic fluid embolism, in pregnancy;
5. Patients whose family members other than the parents and siblings of their offsprings have a history of severe mental illness, such as mental retardation, autism and schizophrenia;
6. Patients undergo acute myocardial infarction in pregnancy;
7. Patients undergo non-spontaneous stroke events due to other causes, such as cerebral infarction or hemorrhage caused by surgery.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ASPP patients and non-ASPP participants during 2010-2024 will be included. For the first part of this study, ASPP patients will be included as cases. This study will also include pregnant or puerperal participants without any history of stroke and non-pregnant or non-puerperal participants with a recent acute stroke event as non-ASPP participants. Non-ASPP participants will be included at Beijing Tiantan Hospital.
  ASPP patients are defined as patients undergo acute stroke events in pregnancy or within 6 weeks postpartum, with the evidence of cerebral infarction or hemorrhage confirmed by neuroimaging corresponding to their symptoms. Considered events will be ischemic stroke, hemorrhagic stroke (including primary and secondary (e.g. due to vascular malformations or systemic disorders) intracerebral hemorrhage and subarachnoid hemorrhage), cerebral venous thrombosis, cerebral artery dissection or central nervous system vasculitis. Transient ischemic stroke will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Long-term modified Ranking Scale scores | At follow-up (assessed between July 2024 to October 2024)
  The modified Ranking Scale (mRS) scores of ASPP and other comparison participants evaluated by specialists. The mRS scores range from 0 to 6, with higher scores indicating worse outcomes.
Recurrent strokes | At follow-up (assessed between July 2024 to October 2024)
  Participants who suffer from recurrent stroke events confirmed by neuroimaging
Apgar scores | At 1 minutes, 5 minutes and 10 minutes after delivery
  Apgar scores of newborns evaluated by specialists. Apgar scores range from 0 to 10, with higher scores indicating better outcomes. Apgar score 8-10 is considered as no asphyxia, 4-7 is considered as mild asphyxia, 0-3 is considered as severe asphyxia.
Age & Stages Questionnaires scores | At follow-up (assessed between July 2024 to October 2024)
  Age & Stages Questionnaires, Third Edition (ASQ-3) scores of offsprings via online self-evaluation. ASQ-3 is divided into 5 subdomains. Scores of each subdomain range from 0 to 60, with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
Short-term modified Ranking Scale scores | At discharge (assessed up to 5 days)
  The modified Ranking Scale (mRS) scores of ASPP and other comparison participants evaluated by specialists. The mRS scores range from 0 to 6, with higher scores indicating worse outcomes.
Strokes during subsequent pregnancies | During subsequent pregnancies (assessed up to 5 days after the 6-week postpartum period of subsequent pregnancies)
  Participants who suffer from stroke events during any subsequent pregnancy
Intrauterine death or stillbirth | Before or at delivery
  Dead fetus in the uterus at any trimester of pregnancy, or birth of a dead infant after 28+1 gestational weeks
Critical illness of offsprings | At follow-up (assessed between July 2024 to October 2024)
  Offsprings requiring hospitalization due to diagnosed diseases within 15 years after birth, including neurological diseases (e.g. epilepsy, cerebral palsy), cardiovascular diseases (e.g. congenital heart disease), gastrointestinal diseases (e.g. necrotizing enterocolitis), respiratory diseases (e.g. allergic asthma), urological diseases (e.g. hypospadias), hematological and immunological diseases and other major diseases

OTHER OUTCOMES:
Length of hospitalization | Between admission and discharge (assessed up to 5 days)
  Time span of hospitalization as a resulting from stroke treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xingju Liu, MD, Principal Investigator — Beijing Tiantan Hospital; Jizong Zhao, MD, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Z, Yin Z, Liu T, Zhang X, Zhang Q, Lu J, Mu L, Dong Y, Liu J, Xiao Y, Chen Y, Song C, Wang Z, Liu Y, Ding W, Zhang L, Shi H, Qi J, Tang B, Wang F, Guo P, Tang Y, Yu M, Zheng W, He Q, Yu J, Zhu A, Fang D, Li G, Bai Y, Zhang Y, Li J, Wang Y, Gao F, Ma Y, Liu Y, Ma L, Yang B, Zhao Y, Ye X, Zhang Q, Zhang Y, Liu X, Zhao J; ASPP Study Group. Clinical characteristics and prognosis of acute stroke in pregnancy and puerperium (ASPP) patients and their offspring: a retrospective, observational, nationwide, multicenter study protocol. Chin Neurosurg J. 2025 Jun 4;11(1):11. doi: 10.1186/s41016-025-00396-5. PMID 40468421